CLINICAL TRIAL: NCT06785025
Title: Women Exercising: Active, and Learning Together for Health (WEALTH) Trial 2.0
Brief Title: Women Exercising, Active, and Learning Together 2.0
Acronym: WEALTH 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRBAM-24-106201
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-01

CONDITIONS: Stress; Depression Secondary to Other Disease; Anxiety; Physical Activity
Keywords: dance; intervention; women; group fitness
MeSH Terms: conditions — Anxiety Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Group 1 will receive access to a 6-week dance fitness intervention (2 classes per week for 30 minutes per class). Group 2 will be a waitlist control condition who will perform their usual routine, but get access to dance fitness classes after all data has been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dance Fitness Group (Experimental): Participants will attend 2 30-minute group-based, dance fitness classes per week for 6 weeks.
  Interventions: Behavioral: Group-Based Dance Fitness Intervention
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will receive no intervention and perform their usual routine. These participants will be given access to dance fitness classes after all data collection has been completed.

INTERVENTIONS:
Behavioral: Group-Based Dance Fitness Intervention — This group-based intervention will be conducted with women only. Women enrolled in the study and assigned to the intervention condition will complete 2 30-minute classes per week for 6 weeks. All classes will be held on a university campus and take place during the lunch hour (12:30-1pm). All classes will be led by a certified group fitness leader who is a member of the research team.
  Arms: Dance Fitness Group

SUMMARY:
The goal of this randomized controlled clinical trial is to determine the efficacy of a 6 week dance fitness intervention has on reducing objective, physiological stress in women between the ages of 30 and 60. It will also learn about its ability to improve mental and psychological health outcomes. The main questions is aims to answer is : 1) To what extent can a 6-week dance fitness intervention improve the health of women? 2) Are intervention effects sustained 4 weeks after the intervention has ended? Researchers will compare the intervention condition to a waitlist control condition. Participants will: 1) complete baseline assessments, 2) complete a six week dance fitness program or complete their usual routine for six weeks, 3) complete immediate post-intervention assessments, and 4) complete follow-up assessments four weeks after the post-intervention assessments.

DETAILED DESCRIPTION:
In the United States, one in five adults (approximately 58 million) is estimated to be living with a mental illness. However, the rate of mental illness is higher in women (27.2%) compared to males (18.1%). High levels of stress, depression, and anxiety are the most reported mental health disorders among women. One protective factor against poor mental health outcomes is participation in physical activity. However, women have been underrepresented in health science studies, precluding us from understanding the best means of promoting physical activity and associated health benefits through intervention.

The Women Exercising, Active, and Learning Together for Health 2.0 (WEALTH 2.0) intervention seeks to understand how a dance fitness intervention may best serve women. This study aims to test the efficacy of a two-arm, group-based physical activity intervention for reducing stress and improving mental health outcomes in midlife women. The two major aims include 1) understanding the immediate- and long-term efficacy of the intervention on physiologic stress and mental health outcomes and 2) determining the associations between change in stress and change in secondary health outcomes. The investigative team will recruit 60 women between the ages of 30 and 60 years to participate in our study. Women will be randomly assigned to an in-person intervention condition or a waitlist control group. Classes will be offered twice per week for 30 minutes for a toal of 6-weeks in the Dance Studio of the Oschner Wellness Center here on the LSU Main Campus by a certified group fitness instructor. Classes will consist of dance fitness content and resistance training exercises to align with the U.S. physical activity guidelines.

The primary outcome of this intervention is physiologically assessed stress (saliva). Secondary outcomes will include perceived stress (questionnaire), depression symptomology (questionnaire), anxiety (questionnaire), body image (questionnaire), social health (questionnaire), intervention adherence (self-report logs), body composition (DEXA scans), and device-measured physical activity (7-day accelerometer protocols). All outcomes will be assessed at three time points: Week 0 (baseline), Week 6 (immediate post-intervention), and Week 10 (follow-up assessment). Achieving the goals of this project will 1) expand upon our previous successful feasibility study, 2) demonstrate the impact of a physical activity intervention and its effect on stress and mental health, 3) better understand the inter-relationships among stress, mental health, and health behaviors/outcomes in midlife women.

ELIGIBILITY:
Inclusion Criteria:

* age 30-60
* body mass index >18
* employed at Louisiana State University
* female

Exclusion Criteria:

* males
* age <18 or >60
* students at Louisiana State University
* Not employed at Louisiana State University
* body mass index <18

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is only including individuals who identify as a female.
Enrollment: 46 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Physiologic Stress | From enrollment to the end of the follow-up period at week 10
  The primary outcome variable of physiologic stress will be assessed through markers in saliva. Samples will be collected using the non-invasive commercially available Salimetrics polyester Oral Swab (SOS) technology (Salimetrics, CA, USA), which has been validated for salivary hormone, sIgA, and alpha-amylase measurements. Immediately after waking up but before getting out of bed, participants will be asked to place one SOS under their tongue for 3 minutes before returning it to the provided vial. Immediately after the first timed saliva collection, participants will be asked to place a second SOS pad under their tongue until full saliva saturation is obtained.

SECONDARY OUTCOMES:
Depression | From enrollment to the end of the follow-up period at week 10
  Secondary outcomes related to depression/sadness will be assessed using the 8-item NIH Toolbox Sadness Short Form. Exemplar items include marking the frequency in the past week for items such as "I felt worthless" or "I felt depressed". This measure uses a five-point scale from "Never" (1) to "Always" (5). This short form has shown both adequate internal consistency α = 0.88) and convergent validity (coefficient = 0.88; compared to the Center for Epidemiologic Studies Depression Scale.
Anxiety | From enrollment to the end of the follow-up period at week 10
  Anxiety will be assessed using the 8-item PROMIS-Anxiety Short Form questionnaire. Exemplar items include marking the frequency in the past week for items such as "I felt uneasy" or "I felt anxious." This measure uses a five-point scale from "Never" (1) to "Always" (5). This measure has demonstrated adequate internal consistency in adult populations (α= 0.93).
Social Health | From enrollment to the end of the follow-up period at week 10
  Social health will be measured using the Emotional Support subscale from the NIH Toolbox Item Bank v3.0 will be used to measure social health. Exemplar items include "I have someone I trust to talk with about my problems" and "I have someone to turn to for suggestions about how to deal with a problem." All items are assessed using a five-point scale with anchors representing frequency in the past month from "Never" (1) to "Always" (5). This measure has demonstrated adequate internal consistency in adult populations (α = 0.97) and construct validity.
Perceived Stress | From enrollment to the end of the follow-up period at week 10
  The secondary outcome of perceived stress will be assessed using the 10-item NIH Toolbox Perceived Stress Survey. Exemplar items include "How often have you felt nervous and 'stressed'?" and "How often have you felt that things were going your way?". All items are assessed using a five-point scale with anchors representing frequency in the past month from "Never" (1) to "Very often" (5). This measure has demonstrated adequate internal consistency in adult populations (α = 0.91).
Body Image | From enrollment to the end of the follow-up period at week 10
  The Multidimensional Body-Self Relations Questionnaire will assess body image. It explores the following constructs: self-esteem, physical fitness, health, concentration on body weight, and concerns about gaining weight. There are 69 items on a scale from 1-5. The higher the score, the greater the satisfaction with body constructs. The following constructs are evaluated in this scale: appearance evaluation, appearance orientation, fitness evaluation, fitness orientation, health evaluation, health orientation, illness orientation, body area satisfaction, overweight preoccupation, and self-classified weight.
Device Measured Physical Activity | From enrollment to the end of the follow-up period at week 10
  Physical activity will be measured with an ActiGraph GT9X Link wrist worn accelerometer worn for 7 days at all times during waking hours. A minimum of 4 days (three weekdays and one weekend day) and a wear time of 10 hours are needed to be included in subsequent analysis. Cut points developed by Montoye et al. will be used to assign sedentary, light, and moderate-to-vigorous physical activity. Participants will receive the accelerometer via the U.S. mail. Written instructions, a QR code for a video demonstration, and contact details of the investigative team will be sent to ensure proper fitting and wearing of the device. The accelerometer will be returned to the research team via prepaid mail envelopes.

OTHER OUTCOMES:
Intervention Compliance | From enrollment to the end of the immediate intervention period at week 6
  Compliance with the intervention will be assessed via attendance logs. For the in-person condition, a research assistant will be present for all classes to report who is in attendance. For the online condition, compliance will be assessed via a self-report log of completing a dance fitness class cross-checked with tracking of participant access and use of the course via the online platform. A continuous variable for total numbers of sessions attended will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Hulteen, PhD, Principal Investigator — Louisiana State University A&M
Locations (1):
- Louisiana State University, School of Kinesiology, Huey P. Long Field House, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing of study info was not approved by IRB